CLINICAL TRIAL: NCT07073300
Title: Endoscopic Findings in Patients Presented With Lower GIT Bleeding in Assiut University Hospitals, a Single-centre Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salah Mohamed Salah Hassan, Resident doctor, Assiut University
Other Study IDs: Endoscopic findings in LGIB
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lower Gastrointestinal Bleeding
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients presented with lower GI bleeding: Patients presented with lower GI bleeding will be investigated with endoscopy to detect different findings
  Interventions: Device: Endoscopy

INTERVENTIONS:
Device: Endoscopy — Upper Endoscopy and colonoscopy will be used

SUMMARY:
Lower gastrointestinal bleeding (LGIB) refers to hematochezia or bright blood passing per rectum of colorectal source distal to ileocecal valve. This differs from the old definition of LGIB which involved small intestine distal to the ligament of Treitz. The new definition of LGIB aligns with current clinical practice and the reality that the majority of LGIB cases come from colorectal origin . In north America, LGIB is one fifth to one third as common as upper gastrointestinal bleeding (UGIB) and represents 30-40 % of all gastrointestinal bleeding cases . 20.5 - 27 cases per 100,000 adults are diagnosed to have LGIB with 21 to 40 cases per 100,000 adults are hospitalized . LGIB has a wide range of aetiologies, presentation and severity. The clinical picture of LGIB depends on patient's age, aetiology and associated comorbidities . Patients can present with overt bleeding in the form of hematochezia which is defined as passage of bright blood per rectum. This should be differentiated from melena (the passage of dark, offensive and digested blood with stool) associated with UGIB . However, 10-15 % of patients with severe acute UGIB can present with hematochezia . In addition, Occult LGIB can present in the form of iron deficiency anaemia or faecal occult bleeding . Causes of LGIB vary significantly according to patient age, lifestyle, dietary habits and geography or race. Some of the most common causes of LGIB include haemorrhoids, colorectal polyps, malignancy, colitis (infective, inflammatory, ischemic, etc.) as well as diverticular disease . However, there are limited data about the common causes of LGIB in upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

* patients with hematochezia and melena. -

Exclusion Criteria:

* poor bowel preparation.
* Inco-operative patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presents with lower gastrointestinal bleeding
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Endoscopic detection of colorectal polyps according to paris classification | Within 24 hours after endoscopy procedure
  Paris Classification of Superficial GI Lesions Main Categories Type 0: Superficial Lesions
  Divided into 3 main types with subtypes:
  1. Type 0-I: Protruded (Polypoid) 0-Ip (Pedunculated): Lesion is on a stalk (like a mushroom). 0-Is (Sessile): Broad-based elevation without a stalk.
  2. Type 0-II: Non-Protruded, Non-Excavated (Flat) 0-IIa (Slightly Elevated): Slight elevation (less than 2.5 mm), often subtle. 0-IIb (Completely Flat): Same level as mucosa, hard to detect without special imaging (e.g., NBI). 0-IIc (Slightly Depressed): A shallow depression; higher risk for malignancy than IIa.
  3. Type 0-III: Excavated (Ulcerated) True ulceration into the mucosa or deeper. Suggests deeper invasion and higher malignancy risk. Combined Morphologies Lesions can be mixed (e.g., 0-IIa + IIc, or 0-Is + IIa).